CLINICAL TRIAL: NCT05437224
Title: A Multicenter Open Label Study to Evaluate Efficacy and Safety of China Made Ambrisentan in Chinese Patients With Pulmonary Arterial Hypertension
Brief Title: Efficacy and Safety Study of Ambrisentan in Chinese Patients With Pulmonary Arterial Hypertension
Acronym: AMBLE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: RenJi Hospital (Other)
Collaborators: Shanghai Zhongshan Hospital (Other); The First Affiliated Hospital with Nanjing Medical University (Other); Shanghai Pulmonary Hospital, Shanghai, China (Other); Xinqiao Hospital of Chongqing (Other); The Affiliated Hospital of Qingdao University (Other); First Affiliated Hospital of Chongqing Medical University (Other); Wuhan Asia Heart Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMBEL
Record Dates: First submitted 2022-06-24; First posted 2022-06-29 (Actual); Last update posted 2022-06-29 (Actual); Status verified 2022-06

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: PAH; ambrisentan
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — ambrisentan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ambrisentan (Experimental): Open Label
  Interventions: Drug: Ambrisentan

INTERVENTIONS:
Drug: Ambrisentan — eligible subjects received 5 mg ambrisentan orally once daily for a 12-week primary evaluation period. Subjects then proceeded to a 12-week dose adjustment period during which dose titration to 10 mg was allowed.

SUMMARY:
This multicenter, open label, single-arm study is aim at investigating the the efficacy and safety of china made ambrisentan in Chinese subjects with PAH.

DETAILED DESCRIPTION:
Pulmonary arterial hypertension is a hemodynamic and pathophysiological state, which can cause progressive hyperplasia of pulmonary vascular walls and elevated pulmonary arterial pressure for various reasons. Ambrisentan is a selective endothelin-A (ETA) receptor antagonist with vasodilatory, antiproliferative and vascular remodeling effects at a dose of 5 mg or 10 mg once daily, oral. A number of international clinical studies have shown that ambrisentan can improve the hemodynamic parameters, WHO functional classification and exercise tolerance of PAH patients, and improve the survival rate. The domestic Ambrisentan tablet is produced by Jiangsu Hansoh Pharmaceutical Group Co., Ltd. under the trade name of "Pu Nuo An". It has been developed and completed according to the consistency evaluation standard after the bioequivalence test, and is currently listed in mainland China. In view of the low price of the domestic ambrisentan, in order to verify its efficacy and safety in the real world, this post-marketing multicenter clinical study was carried out.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old and ≤75 years old, regardless of gender;
* patients weighing ≥ 40 kg;
* Patients diagnosed with PAH in Group 1 of the WHO Updated Clinical Classification of Pulmonary Hypertension (WHO functional class II or III);
* 6 min walk test (6MWT), walking distance ≥ 50 m;
* Right heart catheterization performed within 6 months prior to screening and meeting the following hemodynamic criteria:

  1. mean pulmonary artery pressure ≥ 25 mm Hg；
  2. Pulmonary vascular resistance ≥ 240 dyn·s·cm-5;
  3. Pulmonary artery wedge pressure or left ventricular end-diastolic pressure ≤ 15 mmHg;
* Subject receiving calcium channel blocker (CCB) drugs, only those whose doses have been stabilized for more than 4 weeks at the time of screening are allowed to be included in the study;
* Pulmonary function testing performed within 6 months prior to screening and meeting the following criteria：

  1. Total lung capacity ≥ 60% of normal predicted value;
  2. Forced expiratory volume in one second (FEV1) ≥ 55% of normal expected value;
* Female subjects of childbearing potential must have a negative pregnancy test at the Screening Visit and Day 0;
* Females subjects of childbearing potential must use a medically acceptable method of contraception (eg, hormone therapy, IUD, barrier methods such as condoms or cervical caps) during the study;
* Sign written informed consent

Exclusion Criteria:

* Patients diagnosed with WHO updated PH clinical classification of group 2, 3, 4, 5;
* Endothelin receptor antagonist therapy (eg, bosentan) has been discontinued prior to enrollment due to safety or tolerability concerns (non-drug-induced liver function abnormalities);
* Serum alanine aminotransferase (ALT) or aspartate aminotransferase (AST) levels > 2 times ULN;
* Serum bilirubin level > 1.5 times ULN;
* severe hepatic insufficiency (Child-Pugh class C);
* severe renal insufficiency (creatinine clearance <30 mL/min);
* Hemoglobin concentration < 10 g/dL or hematocrit < 30%;
* Contraindications to treatment identified by laboratory tests, physical examination, medical history, or other investigations
* severe hypotension (diastolic < 50 mm Hg or systolic < 90 mm Hg);
* Clinically significant aortic or mitral valve disease, pericardial constriction, restrictive or congestive cardiomyopathy, fatal arrhythmias, LV ejection fraction < 45%, LV outflow tract obstruction, symptomatic coronary heart disease, spontaneously low blood pressure;
* A history of malignancy within 5 years prior to enrollment, except for basal cell carcinoma of the skin and carcinoma in situ of the cervix;
* Subject taking endothelin receptor antagonists such as ambrisentan, bosentan and macitentan within 4 weeks prior to enrollment;
* pregnant and lactating women;
* Subject deemed unsuitable for participation in this study by other investigators

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2018-12-18 (Actual); Primary Completion 2022-01-09 (Actual); Study Completion 2022-02-06 (Actual)

PRIMARY OUTCOMES:
Change From Baseline to 12 weeks and 24weeks in 6-minute Walk Distance | Baseline, week 12 and week 24
  The 6-minute walk test (6MWT) is a non-encouraged test, performed in a 30 m long flat corridor, where the patient is instructed to walk as far as possible, back and forth around two cones, with the permission to slow down, rest, or stop if needed. These guidelines were provided to all sites. For patients who had never performed a 6MWT previously, a training test was required before the qualifying tests for inclusion were performed.

SECONDARY OUTCOMES:
Time to Clinical Worsening of Pulmonary Arterial Hypertension (PAH) up to Week 24, Assessed as the First Occurrence of a Clinical Worsening Events | From Baseline to week 24
  Clinical Worsening Events included a 15% decrease from baseline on the 6-minute walk test, hospitalization for pulmonary hypertension complications, dosing or escalation of pulmonary hypertension-targeted drugs, atrial septostomy, lung transplantation, or death. Time to clinical worsening of PAH is the time from baseline to the first clinical occurrence of a Clinical Worsening Events.
Change from baseline to week 12 and 24 in Borg Dyspnea Index (BDI) sores | Baseline, week 12 and week 24
  The BDI was calculated by using a 10-point scale (0 = None, 10 = Maximum).
Number of participants with a change from baseline to week 12 and 24 in WHO functional class | Baseline, week 12 and week 24
  The WHO FC was determined by the investigator as follows: Class I - Participants with pulmonary hypertension (PH) but without resulting limitation of physical activity; II- Participants with PH resulting in slight limitation of physical activity; III - Participants with PH resulting in marked limitation of physical activity; IV - Participants with PH with inability to carry out any physical activity without symptoms.
Changes from baseline to week 12 and 24 in BNP plasma levels | Baseline, week 12 and week 24
  BNP is a surrogate maker of heart failure.
Number and severity of Participants With Any Adverse Events | From Baseline to week 24
  An adverse event is defined as any adverse medical event in a patient that is not necessarily causally related to treatment. An adverse event can thus be any adverse or non-therapeutic sign (including abnormal laboratory results), symptom or disease temporally related to the use of the drug product, whether or not considered drug-related.

CONTACTS AND LOCATIONS:
Overall Officials: Jieyan Shen, PhD, Study Chair — Shanghai Jiao Tong University School of Medicine Affiliated Renji Hospital
Locations (1):
- Renji Hospital, Shanghai, China

REFERENCES:
- [Derived] Wang A, Chen M, Zhuang Q, Guan L, Xie W, Wang L, Huang W, Cheng Z, Yu S, Zhou H, Shen J. Time to clinical improvement: an appropriate surrogate endpoint for pulmonary arterial hypertension medication trials. Front Cardiovasc Med. 2023 Jun 12;10:1142721. doi: 10.3389/fcvm.2023.1142721. eCollection 2023. PMID 37378404